CLINICAL TRIAL: NCT00502203
Title: A Phase II Multicenter Trial of Paclitaxel and Carboplatin in Women With Advanced (IIIb, IIIc, IVa and IVb) or Recurrent (All Stages) Malignant Mixed Mullerian Tumors (MMMT) of the Uterus
Brief Title: Paclitaxel and Carboplatin in Women With Malignant Mixed Mullerian Tumors (MMMT) of the Uterus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-229
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Results first posted 2012-01-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2011-12

CONDITIONS: Mixed Tumor, Mullerian
Keywords: Uterine Neoplasms; Endometrial Cancer; Paclitaxel; Taxol; Carboplatin; Paraplatin; Malignant Mixed Mullerian Tumors; MMMT; Immunohistochemical markers
MeSH Terms: conditions — Mixed Tumor, Mullerian; Uterine Neoplasms; Endometrial Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel + Carboplatin (Experimental): Paclitaxel 175 mg/m^2 intravenously (IV) over 3 hours and Carboplatin AUC 5 IV over 1 hour every 21 Days for 6 courses.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — AUC 5 By Vein Over 1 Hour Every 21 Days for 6 Courses
  Other Names: Paraplatin
Drug: Paclitaxel — 175 mg/m^2 By Vein Over 3 Hours Every 21 Days for 6 Courses
  Other Names: Taxol

SUMMARY:
The goal of this clinical research study is to find out if the combination of paclitaxel and carboplatin chemotherapy can shrink or slow the growth of mixed mullerian tumors (MMMT) of the uterus.

DETAILED DESCRIPTION:
Before treatment starts, patients will have a complete check-up, blood tests, a chest x-ray, and a CT scan. Other scans or tests will be done as needed. Women able to have children must have a negative urine pregnancy test. A blood sample will be taken for routine testing once a week during treatment and a month after treatment ends.

Patients will also be asked to complete two questionnaires before they start treatment, before Courses 3 and 5, and at the end of treatment. These questionnaires will help researchers understand how this drug affects patients' daily lives and also identify the side effects caused by this treatment. Each questionnaire will take about 10 minutes to complete.

Patients in this study will be given paclitaxel and carboplatin through a catheter (tube) placed in a vein. Paclitaxel is given first (over 3 hours) followed by carboplatin (over 1 hour). All treatment is given in the outpatient department at M.D. Anderson Cancer Center.

Patients may receive up to 6 courses of treatment. If the disease gets worse or intolerable side effects occur, patients will be taken off study.

-Before each course of treatment, patients will have a checkup. At each checkup, patients will have a physical exam and blood tests. Another CT scan will be done after the third course of treatment. A complete physical exam and a CT scan will also be done at the end of treatment.

This is an investigational study. Both of the study drugs are FDA approved. Their use together in this study is experimental. A total of 50 patients will take part in this multicenter study. About 35 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed advanced (IIIb, IIIc, IVa and IVb) or recurrent (all stages) MMMT.
2. Prior chemotherapy is permitted with the exception of patients previously treated with platinum and/or taxol chemotherapy for this disease.
3. Women of any racial and ethnic group.
4. Eastern Cooperative Oncology Group (ECOG) performance status </= 2.
5. Expected survival of >/= 12 weeks.
6. Patients must have recovered from the side effects of prior therapy (chemotherapy, surgery, or radiation) before entering the study.
7. Adequate liver, renal, and bone marrow function, defined as: a total bilirubin value </= 1.5 mg/dL; serum glutamic pyruvic transaminase (SGPT) </= 2 times upper limit of normal or </= 5 times upper limit of normal when liver metastases are present; serum creatinine </= 1.5 mg/dL; Absolute neutrophil count (ANC) >/= 1,500/ul; platelet count >/= 100,000/ul. All qualifying laboratory parameters must be determined within 1 week prior to first treatment.
8. Participants must agree to practice approved methods of birth control (if applicable).
9. Patients must sign an institutionally approved informed consent.

Exclusion Criteria:

1. Patients with a Zubrod performance status of 3 or greater.
2. Concurrent cancer chemotherapy, radiotherapy or surgery.
3. History of other malignancy (except nonmelanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off all therapy for that disease for a minimum of 5 years.
4. Presence of known untreated brain metastases.
5. Overt psychosis or mental disability or otherwise incompetent to give informed consent.
6. Patients with an active systemic infection.
7. Patients with a serious intercurrent medical illness.
8. Patients with a history of neuropsychiatric or seizure disorders.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2001-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lois M. Ramondetta, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (4):
- United States (4):
  - Loma Linda Cancer Institute, Loma Linda, California
  - MD Anderson Cancer Center, Orlando, Florida
  - Lyndon Baines Johnson Hospital, Houston, Texas
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: August 29, 2001 to May 08, 2009. All recruitment was done at medical clinics.
Period: Overall Study
Arm/Group | Paclitaxel + Carboplatin
Started | 23
Completed | 22
Not Completed | 1
Not completed — Inevaluable | 1

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel + Carboplatin
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 66 [52 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response
Description: Overall response rate including complete (CR) and partial responses (PR) with measurable disease using Response Evaluation Criteria In Solid Tumors (RECIST) assessment. CR: Disappearance of all target and non-target lesions; no evidence of new lesions documented by 2 disease assessments at least 4 weeks apart. PR: At least 30% decrease in sum of longest dimensions (LD) of all target measurable lesions reference baseline sum of LD; no unequivocal progression of non-target lesions and no new lesions. Documentation by 2 disease assessments at least 4 weeks apart is required.
Time Frame: 24 Months
Population: Thirteen participants had measurable disease therefore evaluable for a complete or partial response.
Measure: Number; unit: participants
Arm/Group | Paclitaxel + Carboplatin
Number analyzed (Participants) | 13
participants | 8

ADVERSE EVENTS:
Time Frame: 7 years and 11 months
Arm/Group | Paclitaxel + Carboplatin
Serious Adverse Events (participants affected / at risk) | 9/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel + Carboplatin (N=23)
Neutropenia (Blood and lymphatic system disorders) | 9
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel + Carboplatin (N=23)
Allergic Reaction (General disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 23
Anemia (Blood and lymphatic system disorders) | 9
Anorexia (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 21
Headache (General disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Infection (Infections and infestations) | 1
Neuropathy (sensory) (Nervous system disorders) | 14
Neuropathy (hearing) (Nervous system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 11
Neutropenic Fever (Blood and lymphatic system disorders) | 3
Mucositis (Gastrointestinal disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 15
Nausea (Gastrointestinal disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Vomiting (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No